CLINICAL TRIAL: NCT07351448
Title: Research on the Extraction of Tongue and Facial Diagnosis Features of Psoriasis Vulgaris in Traditional Chinese Medicine and Its Correlation With Laboratory Indicators
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-206
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis (PsO); Traditional Chinese Medicine (TCM); Diagnosis
MeSH Terms: conditions — Psoriasis; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — The collected sample is venous blood.The volume collected for each patient is 8 mL. After centrifugation, the serum is extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-psoriasis subjects: Who visit for non-psoriasis skin conditions such as eczema or acne, and have been professionallyand confirmed by doctors not to have psoriasis, will be chosen as the Non-psoriasis subjects.
  Interventions: Other: No intervention
- Psoriasis blood stasis syndrome group: Patients with psoriasis diagnosed as having blood stasis syndrome
  Interventions: Other: No intervention
- Psoriasis non-blood stasis syndrome group: Patients with psoriasis diagnosed as not having blood stasis syndrome
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, no intervention implemented.

SUMMARY:
Psoriasis Vulgaris is a chronic, inflammatory, and immune-activated skin disease. It is the most common type of psoriasis, accounting for approximately 85-90% of all psoriasis patients. Its clinical features include erythema, papules, covered with varying scales, a long course of disease, and recurrent attacks. According to traditional Chinese medicine, psoriasis is mainly characterized by blood heat syndrome, blood stasis syndrome and blood dryness syndrome, accounting for more than 90% of all syndrome types. The TCM syndrome differentiation and treatment of psoriasis also attach great importance to the transformation and evolution of TCM syndrome types. For instance, the three syndrome types of blood heat syndrome, blood stasis syndrome and blood dryness syndrome are not static and can transform into each other. For example, blood heat syndrome can develop into blood dryness syndrome as the disease progresses, blood dryness syndrome can transform into blood stasis syndrome, and blood stasis syndrome can also transform into blood heat syndrome or blood dryness syndrome. Observation is an important diagnostic method in traditional Chinese medicine. The images of tongue and face diagnosis contain a lot of important clinical information. They can objectively reflect the prosperity and decline of qi and blood in the human body, the nature of diseases, the depth of the lesion location, the prognosis of the disease, and can also reflect the physiological and pathological changes of the body. In recent years, significant progress has been made in the research of digital and intelligent technologies for tongue and facial diagnosis. Introducing objective indicators such as tongue diagnosis, facial diagnosis and pulse diagnosis into the evaluation research of diseases has become a hot topic. This project, by analyzing the clinical tongue and facial image data of patients with psoriasis vulgaris and combining it with clinical laboratory indicators, fuses and analyzes the characteristic parameters of patients' tongue and facial diagnosis with blood biochemical indicators, metabolomics and other data. This is helpful to reveal the disease occurrence pattern of patients with blood stasis type psoriasis and construct a diagnostic model for blood stasis syndrome of psoriasis. At the same time, it provides a powerful decision support tool for clinical practice and also helps deepen our understanding of the complex process of the occurrence of blood stasis type psoriasis, thereby providing a solid scientific basis for formulating precise diagnostic and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the non-psoriasis subjects: (1) Those who do not meet the Western medical diagnostic criteria for psoriasis; （2) No gender restrictions; 18 years old ≤ age ≤ 65 years old; (3) Understand and agree to participate in this study and sign the informed consent form; Inclusion criteria for the psoriasis blood stasis syndrome group: (1) Those who meet the Western medical diagnostic criteria for psoriasis and whose TCM syndrome classification belongs to blood stasis syndrome; (2) No gender restrictions; 18 years old ≤ age ≤ 65 years old; (3) Understand and agree to participate in this study and sign the informed consent form.

Inclusion criteria for the psoriasis non-blood stasis syndrome group: (1) Those who meet the Western medical diagnostic criteria for psoriasis and whose TCM syndrome classification belongs to blood heat syndrome/blood dryness syndrome; (2) No gender restrictions; 18 years old ≤ age ≤ 65 years old; (3) Understand and agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* (1) Due to various reasons, the collected tongue and facial images may be unclear or cannot be successfully monitored and analyzed; (2) For those subjects whose facial makeup or tongue coating is applied, the information obtained from tongue and facial diagnosis may be inaccurate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study intends to select 150 patients with blood stasis syndrome of psoriasis who visited the Department of Dermatology of Yueyang Integrated Traditional Chinese and Western Medicine Hospital affiliated to Shanghai University of Traditional Chinese Medicine, as well as 150 patients with non-blood stasis syndrome of psoriasis. Additionally, 150 people who visited the hospital due to non-papular psoriasis skin diseases such as eczema or acne, and who were confirmed by professional doctors to have no psoriasis, will be selected as the non-psoriasis subjects.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Images | 1 day (Collect the images of the patient's tongue and face using a tongue surface scanner)

SECONDARY OUTCOMES:
Serum metabolomics data | 1 day (Collect the serum and send it to the testing company for metabolomics testing)
Psoriasis Area and Severity Index (PASI) | The researcher conducted a Psoriasis Area and Severity Index (PASI) assessment on the psoria on the 1 day of sample collection
Inflammatory factor | 1 day （Collect serum and test the levels of IFN-γ, TNF-α and IL-17）

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China